CLINICAL TRIAL: NCT02597166
Title: The Effects of Anti-Viral Therapy on the Clinical Status, Quality of Life, and Survival of Patients With Decompensated Cirrhosis Due to Hepatitis C Genotype 1 Infection
Brief Title: Effects of Harvoni in Patients With Decompensated Cirrhosis Due to Hepatitis C Genotype 1 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Florence Wong, MD, Hepatologist, Professor Division of Gastroenterology, Department of Medicine University of Toronto, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-CA-337-1960
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Hepatitis C, Chronic; Cirrhosis, Decompensated
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ledipasvir/Sofosbuvir (Other): Each tablet contains 90 mg ledipasvir and 400 mg sofosbuvir, given orally, once daily for 24 weeks.
  Interventions: Drug: Ledipasvir/Sofosbuvir

INTERVENTIONS:
Drug: Ledipasvir/Sofosbuvir — Each tablet of Harvoni contains 90 mg ledipasvir and 400 mg sofosbuvir.
  Other Names: Harvoni

SUMMARY:
There are now several licensed drug treatments for patients with HCV infection. These medications have been shown to be very effective in getting rid of the virus in patients with HCV infection including those with early stages of cirrhosis without complications known as compensated cirrhosis, with a greater than 90% cure rate. At present, there are very little data to show that treating patients with HCV infection and decompensated cirrhosis will give the same effects. However, patients with decompensated cirrhosis as a result of hepatitis B infection who received treatment to control their virus show improvement of their overall liver condition, and the liver complications of many of these patients disappeared. Also, patients with cirrhosis due to excess alcohol and who stopped drinking also showed improvement in liver function and their complications of cirrhosis coming under control. Therefore, treatment of patients with HCV infection and decompensated cirrhosis is expected to show the same positive effects, because the underlying cause of cirrhosis is coming under control. Harvoni is a combination of two direct-acting antivirals (ledipasvir and sofosbuvir) that prevents the hepatitis C virus from copying and multiplying themselves, allowing the body to clear the virus from their systems and be cured of HCV infection. This study is being conducted to find out if treatment with Harvoni will lead to clearance of HCV infection in patients with decompensated cirrhosis giving rise to improvement in liver function, together with improvement of quality of life and survival.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is one of the most common causes of liver cirrhosis worldwide. The progression of liver cirrhosis can lead to a myriad of complications including ascites, variceal bleeding, hepatic encephalopathy, hepatorenal syndrome, and hepatocellular carcinoma. The development of these complications or decompensation can lead to a dismal survival of 50% at 6 months, especially if the underlying cause of the liver cirrhosis is not treated. The cost of caring for these patients with decompensated cirrhosis is extremely high. Despite this, every effort is being made to maintain these patients in reasonable health until liver transplant becomes available for them. Yet these patients continue to have poor quality of life because of the various symptoms related to decompensated cirrhosis, and spend much time visiting health care facilities for both outpatient and inpatient care.

The recent availability of potent and effective anti-viral therapy has revolutionized the management of patients with hepatitis C infection. With a >90% cure rate, many patients with compensated cirrhosis, once treated, will not progress further to develop decompensation. With the passage of time, the liver cirrhosis may even regress to a non-cirrhotic state. Published data on treatment of decompensated cirrhosis with hepatitis C infection is still scanty. However, patients with decompensated cirrhosis due to hepatitis B infection who received effective anti-viral therapy not only improved their overall clinical status, many of these patients reverted from a decompensated to a compensated state, associated with improved survival. Likewise, patients with alcoholic cirrhosis who abstain from alcohol will also have improvement in liver function and reduction in complications of cirrhosis. Therefore, treatment of decompensated cirrhotic patients with hepatitis C is expected to show the same beneficial effects, because the underlying cause of cirrhosis is coming under control.

The primary objective of this study is to assess the effects of anti-viral therapy on the clinical status, quality of life and survival of patients with decompensated cirrhosis due to chronic hepatitis C genotype 1 infection.

After completion of all initial investigations, patients will be started on Harvoni 90 mg ledipasvir/400 mg sofosbuvir (one tablet) daily. The course of treatment will be 24 weeks. Patients will be reviewed at monthly intervals as per standard of care. At each clinic visit, patients with have blood tests including complete blood count, renal function, electrolytes, liver enzyme and liver function tests, HCV RNA will be done at week 4, week 12, week 24 during treatment, and then again at week 12 post completion of treatment. Annual ultrasounds and surveillance gastroscopies will be organized as per standard of care.

Patient will be followed for 1 year post completion of treatment, and have repeat quality of life questionnaires at end of treatment, and thereafter at 6 and 12 months. Patients will also be monitored for the development of further complications of cirrhosis (if any), hospital admissions, reasons for hospital admissions, lengths of hospital stays, survival, and liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

Treatment-naïve and treatment-experienced patients with CHC genotype 1 infection and decompensated cirrhosis as defined by one of the following:

* history of variceal bleeding
* presence or history of ascites
* history of grade III-IV hepatic encephalopathy
* Coagulopathy with an INR>1.7
* Jaundice with a serum bilirubin of >85µmol/L

Cirrhosis is defined as any one of the following:

* A liver biopsy performed prior to the study showing cirrhosis (F4)
* Fibroscan performed within 12 calendar months of the start of this study with a result of > 12.5 kPa
* A Fibrotest ® score of >0.75

Exclusion Criteria:

* Patients older than 75 years
* Presence of hepatoma at entry
* Patients awaiting living-related liver transplantation
* MELD score of >30
* Significant co-morbid condition(s) with a life expectancy of <6 months
* HIV co-infection
* HBV co-infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Improvement of quality of life based on Chronic Liver Disease Questionnaire | one year
  Improvement of quality of life based on Chronic Liver Disease Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Florence Wong, MD, Principal Investigator — University Health Network - Toronto General Hospital
Locations (1):
- University Health Network - Toronto General Hospital, Toronto, Ontario, Canada